CLINICAL TRIAL: NCT07368101
Title: Outcome of Chronic Subdural Hematoma: Double Burr Hole Versus Single Burr Hole With Subdural Drain Evacuation
Brief Title: Outcome of Chronic Subdural Hematoma Management With Double Burr Hole Craniotomy Versus Single Burr Hole Craniotomy and Subdural Drain Evacuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Muhammad Hassan tabish, Muhammad Hassan Tabish , MBBS, Neurosurgery Resident / Principal Investigator, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2024/1395/SIMS
Record Dates: First submitted 2026-01-12; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double burr Hole Arm (Experimental): this arm includes patient who receive double burr hole craniotomy surgical procedure for drainage of chronic subdural hematoma
  Interventions: Procedure: Double Burr hole Craniotomy
- Single Burr Hole Arm (Experimental): this arm includes patient who receive single burr hole craniotomy surgical procedure for drainage of chronic subdural hematoma
  Interventions: Procedure: Single Burr hole Craniotomy

INTERVENTIONS:
Procedure: Single Burr hole Craniotomy — Single Burr hole made at the point of highest collection of hematoma in subdural space in brain.
  Arms: Single Burr Hole Arm
Procedure: Double Burr hole Craniotomy — Two burr hole made in skull each at parietal eminence and around superior temporal line to drain chronic subdural hematoma
  Arms: Double burr Hole Arm

SUMMARY:
The goal of this clinical trial is to compare the outcome of double burr hole versus single burr hole in patients of chronic subdural hematoma undergoing subdural drain evacuation.

The main questions it aims to answers are

1. Which one of the surgical method i.e single burr hole or double burr hole is clinically superior with better post operative prognosis for the drainage of chronic subdural hematoma.

2 Compare the post operative complications in both the techniques in term of wound infection hospital stay duration , recurrence and mortality.

participants will be divided in two groups one group will be treated with single burr hole technique second group will be treated with double burr hole technique.

After procedure, patients will be followed-up in hospital until discharge and total hospital stay will be noted. Patients will be followed-up further in OPD . During follow-up, patients will be evaluated for wound infection, recurrence and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-70 years both genders diagnosed with subdural hematoma

Exclusion Criteria:

* • Patients in shock (BP≤100/60 mmHg) or history of seizures

  * Patients with bleeding disorder (PT>15 sec) or intake of anti-coagulants
  * Patients undergoing or already had ventriculoperitoneal shunt
  * Patients with epilepsy, or obsessive compulsive decoder
  * Patients with already operated for subdural hematoma
  * Patients with post-cerebrospinal fluid diversion subdural hematoma

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Recurrence Of Chronic Subdural Hematoma | From date of surgery until radiologically confirmed recurrence (defined as subdural hematoma volume >15 mL or significant mass effect on CT brain) requiring repeat intervention, assessed up to 3 months postoperatively
  recurrence rate of chronic subdural hematoma evaluated if volume of sdh >15ml or significant mass effect on CT brain within 3 months post operatively
quantity of hematoma evacuated | Measured intraoperatively at the time of surgery and cumulatively measured postoperatively from surgery until removal of the subdural drain, assessed up to 72 hours postoperatively.
  Intraoperatively evacuated hematoma quantity measured in millilitres and also includes the quantity obtained in subdural drain till 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan Tabish, MBBS, Principal Investigator — Services Hospital / Services Institute of Medical Sciences
Locations (1):
- Services Institute of Medical Sciences / Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No